CLINICAL TRIAL: NCT03524573
Title: Delayed vs. Early Laparoscopic Appendectomy : A Randomized Controlled Trial (The DELAY Trial)
Brief Title: (D)Elayed vs. (E)Arly (L)Aparoscopic (A)Ppendectom(Y)
Acronym: DELAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Sunil Patel, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SURG-402-17
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Appendectomy (Experimental): Patients will undergo appendectomy the morning following the decision to operate. This group will have an anticipated delay between 3 - 14 hours from the decision to operate, with a surgical start time between 0530 - 0900.
  Interventions: Procedure: Appendectomy
- Immediate Appendectomy (Active Comparator): Patients will undergo appendectomy within 6 hours of the decision to operate. Surgery will take place between 2000 - 0400.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Appendectomy is the surgical removal of the appendix.

SUMMARY:
The DELAY Trial will compare immediate (< 6 hours from decision to operate) to delayed (Surgery to take place the following morning) appendectomy in adult patients presenting to the emergency department with suspected acute appendicitis. The primary outcome will be 30 day postoperative complications.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to assess the effect of timing of surgery on surgical complications in patients undergoing appendectomy for acute appendicitis at one of two participating institutions.

Early appendectomy in patients diagnosed with acute appendicitis has been a mainstay of treatment. Timely intervention is recommended to avoid the risks associated with perforated appendicitis, which has been shown to increase the risk of post-operative complications compared to non-perforated appendicitis. However, some studies have suggested that delaying appendectomy does not increase complications. Several studies have also assessed the safety of nighttime operating with conflicting results. Some suggest that delaying surgery until daytime is safe.

This study is a prospective, randomized controlled trial with blinding of the outcome assessors. Eligible participants will be adult patients diagnosed with acute appendicitis with an expected operative start time between 2000-0400. Patients randomized to the intervention group will have delayed surgery after 0530 the following morning to avoid nighttime operating. Patients randomized to the control group will receive immediate surgery within 6 hours of the decision to operate. The follow up period will be a minimum of 30 days. Independent outcome assessors will assess patients during their postoperative course in hospital as well as in the outpatient follow up clinic.

The primary outcome for this study is complication occurring within 30 days of surgery. Complication includes any of the following: mortality, readmission to hospital, emergency department (ED) visit, percutaneous drain insertion, reoperation, prolonged hospital stay greater than 7 days, and a predefined list of postoperative complications. Secondary outcomes include perforated appendicitis, operative time, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age
* Imaging confirmed diagnosis of appendicitis (ultrasound or CT or MRI)
* Expected time of operation between 2200 - 0400 and occurs within 6 hours of the decision to operate

Exclusion Criteria:

* Patients with hemodynamic instability
* Patients with suspected sepsis
* Unknown diagnosis
* Presence of abscess on CT Scan
* Diagnosis of missed appendicitis
* Pregnancy
* Patients who are not surgical candidates
* Patients who are not competent to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
30 Day Post Operative Complications | within 30 days of surgery

SECONDARY OUTCOMES:
Perforated Appendicitis | At time of surgery
Operative Time | At time of surgery
Length of Stay - Index Admission | Index Admission
Length of Stay - Index admission plus any additional admissions within 30 days of surgery | 30 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patel SV, Zhang L, Mir ZM, Lemke M, Leeper WR, Allen LJ, Walser E, Vogt K. Delayed Versus Early Laparoscopic Appendectomy for Adult Patients With Acute Appendicitis: A Randomized Controlled Trial. Ann Surg. 2024 Jan 1;279(1):88-93. doi: 10.1097/SLA.0000000000005996. Epub 2023 Jul 13. PMID 37436871